CLINICAL TRIAL: NCT00363038
Title: Effects of Topical Vitamin K, Vitamin K and Retinol, and Arnica on Post-Laser Bruising
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Northwestern University (Other)
Responsible Party: Principal Investigator, Murad Alam, Associate Professor of Dermatology, Northwestern University
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 1253-015
Record Dates: First submitted 2006-08-10; First posted 2006-08-15 (Estimated); Results first posted 2012-12-04 (Estimated); Last update posted 2021-12-03 (Actual); Status verified 2021-12

CONDITIONS: Ecchymosis
Keywords: Bruising; Topical 20% arnica
MeSH Terms: conditions — Ecchymosis; Contusions | interventions — Vitamin K

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (1):
- Bruising (Experimental): Bruises at three time points: immediate after bruise creating, and at 1 and 2 weeks.
  Interventions: Drug: Petrolatum United States Pharmacopeia (USP); Drug: Vitamin K and retinol ointment; Drug: Arnica ointment; Drug: Vitamin K ointment

INTERVENTIONS:
Drug: Petrolatum United States Pharmacopeia (USP) — Topical formation applied to bruise twice daily for 2 weeks.
Drug: Vitamin K and retinol ointment — Topical formation applied to bruise twice daily for 2 weeks.
Drug: Arnica ointment — Topical formation applied to bruise twice daily for 2 weeks.
Drug: Vitamin K ointment — Topical formation applied to bruise twice daily for 2 weeks.

SUMMARY:
The objective of this study is to assess the comparative utility of topical formulations in hastening the resolution of skin bruising. For each subject, four standard bruises of 7 mm diameter each were created on the bilateral upper inner arms, 5 cm apart, two per arm, using a 595-nm pulsed-dye laser. Randomization was used to assign one topical agent (5% vitamin K, 1% vitamin K and 0.3% retinol, 20% arnica or white petrolatum) to exactly one bruise per subject, which was then treated under occlusion twice a day for 2 weeks. A dermatologist rated bruises in standardized photographs immediately after bruise creation and at week 2.

ELIGIBILITY:
Inclusion Criteria:

* Age 20-60
* Subjects are in good health.
* Subjects have willingness and the ability to understand and provide informed consent for participation in the study.

Exclusion Criteria:

* Subjects who are currently using any anticoagulation therapy (Warfarin, Heparin, Aspirin)
* Subjects who have a history of bleeding disorders.
* Subjects who are unable to understand the protocol or to give informed consent
* Subjects with mental illness
* Subjects who are pregnant or nursing.
* Subjects who have active systemic or local infection
* Subjects with systemic or local skin disease.
* Subjects with systemic illness.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2006-07; Primary Completion 2006-08 (Actual); Study Completion 2006-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Murad Alam, MD, Principal Investigator — Northwestern University
Locations (1):
- Northwestern University Feinberg School of Medicine, Department of Dermatology, Chicago, Illinois, United States

REFERENCES:
- [Background] Leu S, Havey J, White LE, Martin N, Yoo SS, Rademaker AW, Alam M. Accelerated resolution of laser-induced bruising with topical 20% arnica: a rater-blinded randomized controlled trial. Br J Dermatol. 2010 Sep;163(3):557-63. doi: 10.1111/j.1365-2133.2010.09813.x. PMID 20412090

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited at a university-based dermatology department in an urban center.
Groups:
- Average Bruise Improvement: pulsed dye laser induced four 1 cm bruises at least 5 cm apart on the skin of the upper arm (two bruises on each arm). Subjects applied different topical ointments on each of their bruises twice a day. Ointments were: 5% vitamin K cream; 1% vitamin K and 0.3% retinol cream; 20% topical arnica; white petrolatum United States Pharmacopeia (USP) as placebo.
Period: Overall Study
Arm/Group | Average Bruise Improvement
Started | 16
Completed | 16
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Average Bruise Improvement: pulsed dye laser induced four 1 cm bruises at least 5 cm apart on the skin of the upper arm (two bruises on each arm). Subjects applied different topical ointments on each of their bruises twice a day. Ointments were: 5% vitamin K cream; 1% vitamin K and 0.3% retinol cream; 20% topical arnica; white petrolatum USP as placebo.
Arm/Group | Average Bruise Improvement
Number analyzed (Participants) | 16
Age, Continuous [Mean (Full Range); unit: years] | 26 [21 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 6
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Average Bruise Change
Description: Mean change in bruising level detected by dermatologist rater on Visual Analogue Scale at 2 weeks compared with baseline for each of the four agents (Petrolatum USP, Vitamin K and retinol ointment, Vitamin K ointment, Arnica ointment). When responding to a VAS item, respondents specify the bruise severity by indicating a position along a continuous line between two end-points (0 and 10, 10 being the most bruised).
Time Frame: Baseline and 2 weeks
Measure: Mean (Standard Deviation); unit: Units on a Scale
Arm/Group | Average Bruise Improvement
Number analyzed (Participants) | 16
Units on a Scale
  Petrolatum USP | -3.68 (0.68) [-10 to 10]
  Vitamin K and retinol ointment | -3.71 (0.60) [-10 to 10]
  Vitamin K ointment | -3.88 (0.71) [-10 to 10]
  Arnica ointment | -4.13 (0.84) [-10 to 10]

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Average Bruise Improvement
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 5/16
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Average Bruise Improvement (N=16)
Redness and swelling at the treated sites (Skin and subcutaneous tissue disorders) | 4 (4)
Blistering (Skin and subcutaneous tissue disorders) | 1 (1)

LIMITATIONS AND CAVEATS:
As only laser-induced bruising on the inner arm was studied, it remains to be seen if this result can be generalized to other postoperative bruises and at other anatomical sites.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No